CLINICAL TRIAL: NCT01619904
Title: Effects of Goal-Directed Therapy on Inflammatory Mediators and Postoperative Outcome in Pancreas Transplant: a Prospective Randomised Clinical Trial
Brief Title: GDT Vs ST for Pancreas Transplant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Hussein Khambalia, Senior Clinical Research Fellow, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAK 14
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Pancreas Transplantation
Keywords: Pancreas Transplantation; Goal-directed therapy; Outcomes; Immunometric
MeSH Terms: interventions — Early Goal-Directed Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal-Directed Therapy (Experimental)
  Interventions: Procedure: Goal-Directed Therapy
- Standard Therapy (Active Comparator)
  Interventions: Procedure: Standard Therapy

INTERVENTIONS:
Procedure: Goal-Directed Therapy — Peri-operative optimisation of fluid status, based on Oxygen Delivery
  Arms: Goal-Directed Therapy
Procedure: Standard Therapy — Following standard protocol during peri-operative period
  Arms: Standard Therapy

SUMMARY:
A Pancreas Transplant is the accepted treatment in patients with Insulin Dependent Diabetes Mellitus (IDDM) and end-organ failure. Simultaneous Pancreas and Kidney (SPK) Transplant is done in over 90% of cases. At present there is a 5- 8% 30-day mortality with over 80% graft survival at 1 year. At Manchester Royal Infirmary (MRI) approximately 40 cases are done per year.

Goal-Directed Therapy (GDT) involves fluid resuscitation intra-operatively and early in the post-operative period, guided by cardiac output monitoring. The mechanism of therapeutic benefit is thought to be related to improved tissue oxygenation and oxygen delivery. There are a number of studies showing significantly improved biochemical markers of inflammation in animal models and in studies on septic patients (patients with an overwhelming infection) following GDT. Studies have also shown that GDT improves clinical outcome in post-operative patients and in serum inflammatory mediators. These studies have looked at "major abdominal surgery" but none have investigated transplant patients. Given the nature of surgery we feel that our patients would benefit with reduced Intensive Care Unit stay, reduced length of hospital stays and reduced rates of post-operative complications.

The study will be conducted on all adult patients undergoing pancreas transplant at MRI. It will last for 2 years and we hope to recruit 60 patients

Patients will be randomised into Standard Therapy (ST) or GDT groups, with ST being current practice. Each intervention will last for six hours post-operatively before continuing with normal care thereafter. Omental fat biopsies will be taken from patients intra-operatively and blood samples will be taken from patients at regular intervals for 72 hours intra- and post- operatively. Patients will be followed up daily while an in-patient and at three-monthly intervals in out-patients for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All adult pancreas transplant recipients between November 2011- November 2013

Exclusion Criteria:

* Those unable to consent
* Paediatric recipients
* Patients unable to meet follow-up protocol
* Patients with a contra-indication to central venous catheterisation
* Patients with advanced directives, restricting the implementation of the study protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | 2 years

SECONDARY OUTCOMES:
Inflammatory marker levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Khambalia, BMBS, Principal Investigator — CMFT, University of Manchester
Locations (1):
- Manchester Royal Infirmary, Manchester, Manchester, United Kingdom